CLINICAL TRIAL: NCT05613530
Title: Mobile Application (Max NEONAT) as a Clinical Support Tool for Neonatal Resuscitation in the Delivery Room: A Simulation-based Bicentric Randomized Controlled Trial.
Brief Title: Mobile Application as a Clinical Decision Support Tool for Neonatal Resuscitation in the Delivery Room
Acronym: MAXnéonat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Study Director, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MAX néonat
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Simulation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital MAX néonat (intervention group or " MAX + group") (Experimental): Participants use a digital, hand-held, cognitive aid (a mobile application named "MAX NEONAT") and the ILCOR 2020 algorithm poster.
  This group consists of a resident in pediatrics + 2 midwifes.
  Interventions: Behavioral: MAX NEONAT
- MAX néonat on poster/paper (control group or " MAX - group") (Active Comparator): Participants have no cognitive aid
  Interventions: Behavioral: standard of care

INTERVENTIONS:
Behavioral: MAX NEONAT — Participants use a digital, hand-held, cognitive aid (a mobile application named "MAX NEONAT") and the ILCOR 2020 algorithm poster.
  This group consists of a resident in pediatrics + 2 midwifes.
  Arms: digital MAX néonat (intervention group or " MAX + group")
Behavioral: standard of care — no cognitive aid but poster/paper only
  Arms: MAX néonat on poster/paper (control group or " MAX - group")

SUMMARY:
The need for neonatal cardiopulmonary resuscitation in the delivery room is rare with less than 1% of newborns requiring advanced resuscitation. The use of clinical decision support tools to guide practitioners on medical procedure steps is recognized by the medical community. In this randomized bi-centric controlled study, we investigate the effect of a mobile phone application on technical and non-technical performance of student trinomials managing simulated critical neonatal events

DETAILED DESCRIPTION:
The need for neonatal cardiopulmonary resuscitation in the delivery room is rare with less than 1% of newborns requiring advanced resuscitation: Approximately 85% of babies born at term will initiate breathing spontaneously at birth. An additional 10% will do so in response to stimulation and drying. However, approximately 5% of term infants receive positive-pressure ventilation to successfully transition, 2% are intubated, 0.1% receive cardiac compressions, and 0.05% receive compressions with Epinephrine. These events are rare but stressful and require fast response. High stress impairs cognitive skills, including decision making, short-term memory, knowledge recall, and situational attention. In order to help practitioners, guidelines and algorithm exists: The neonatal resuscitation program (NRP) and International Liaison Committee on Resuscitation (ILCOR) algorithm outlines essential steps to take to assist a neonate immediately after birth. ILCOR algorithm poster is present in every delivery room in France. Nevertheless, studies have shown a 16-55% error rate in adherence to the NRP algorithm. Despite periodic training skills deterioration, technical performance, and aptitude to follow recommendations decline over time.

The use of cognitive aids might be a solution to prevent errors in critical situation. Cognitive aids are defined as "prompts designed to help users complete a task or series of tasks." The design of cognitive aids includes posters, checklists, mnemonics, or digital tools like computer programs or smartphone applications. Poster or checklist cognitive aids are widely used to help health care to follow standardized procedures while facing high-cognitive loads situations. Many digital cognitive aids have been developed in intensive care (cardiac arrest) and anesthesiology both in adult and pediatric fields. They have been shown to improve technical skills along with guideline adherence in adult's study. Influence of cognitive aids on technical and nontechnical skills has not been investigated extensively and is still controversial in pediatrics. In neonatology some studies exist but with discordant results. MAX (Medical Assistance eXpert) is a mobile French cognitive aid available on smartphone or tablet. The use of MAX has been shown to improve technical and nontechnical skill in previous adult studies. To evaluate the usefulness of digital cognitive aid in neonatal critical situations, ILCOR 2020 algorithm was included in MAX. A previous unpublished pilot study in neonatal simulated cardiopulmonary arrest shown feasibility in trinomials and improvement in technical skill.

We performed an unblinded randomized trial comparing the use of a digital, hand-held, cognitive aid (a mobile application named "MAX NEONAT") and the ILCOR 2020 algorithm poster, vs. without cognitive aid, to test the hypothesis that MAX NEONAT could improve technical performance and affect non-technical performance of pediatric residents and mid wife-students facing simulated neonatal cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric residents in Lyon and Caen University with at least a three-month clinical experience in a neonatal intensive care unit and one or more high fidelity neonatal resuscitation simulation sessions participation
* All midwife students in Lyon and Caen which had benefited from teaching classes on neonatal resuscitation

Exclusion Criteria:

* Participants who didn't attend one of the scheduled study sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a technical performance score, adapted from of a previously published checklist score. The technical score follows the (International Liaison Committee on Resuscitation recommendations (ILCOR). | DAY 1
  the NRP checklist ( Neonatal Rescucitation Program) score we utilized is a previously published technical performance score adapted from the ILCOR 2020 recommendations. This revised NRP score is composed of 27 points. For each action, trinomials are given a score of 0 for not performing the action, 1 for performing the task correctly and in order.

SECONDARY OUTCOMES:
non-technical skills | Day 1
  non-technical skills, evaluated by an adaptation of a previously published checklist score. The non-technical score includes three categories: leadership, teamwork and task management. The score has a total of 36 points. A questionnaire evaluating the functionality and usefulness of the mobile phone application will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Beissel, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- CHU LYON, Lyon, France